CLINICAL TRIAL: NCT03784911
Title: Assessment of Body Composition During Cancer Treatment Using the SOZO Device
Brief Title: Body Composition During Cancer Treatment
Acronym: DuringSOZO
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Collaborators: ImpediMed Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00077264
Record Dates: First submitted 2018-08-08; First posted 2018-12-24 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: Body Composition; SOZO; Cancer; Cancer Treatment; Impedimed
MeSH Terms: conditions — Neoplasms | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- During Cancer Treatment Group: Participants' body composition will be estimated using a SOZO device at 5 different time points across their cancer treatment. Participant will also complete questionnaires and physical assessments during each study visit. These include waist & hip measurements, weight/BMI, brief fatigue inventory, timed up and go test, cancer distress assessment, ECOG performance status, hand grip strength test, and 24-hour food recall. DEXA scans will be performed before treatment and after completion of treatment.
  Interventions: Device: SOZO Device; Device: DEXA Scan

INTERVENTIONS:
Device: SOZO Device — SOZO device will estimate fluid status, total body composition, metabolic report, skeletal muscle mass, phase angle, body mass index, weight, and hydration index analysis. SOZO measurements will be performed before the start of cancer treatment, at the 1/4, 1/2, and 3/4 time points of treatment, and after completion of treatment. Participants be asked to fast for at least 8 hours before each visit, but water may be consumed to ensure they are well-hydrated. Participants will be asked to provide a urine sample at each visit and to report the color of your urine to the staff so they can determine how well hydrated the participants are. If not hydrated to the extent needed, participants will be asked to drink water and repeat the urine sample again after 30 minutes.
Device: DEXA Scan — DEXA scan bone density reading with hip and spine measurements as well as a whole body composition scan will be performed. Where DEXA cannot be collected on the same day as other study assessments, Weight/BMI, Urine Color, and SOZO should all be collected (or repeated if already done) to coincide with the DEXA scan if SOZO is available at DEXA location.

SUMMARY:
The purpose of this study is to assess how bone density and body composition changes over a cancer patient's treatment via SOZO measurements, DEXA scan (bone density and whole body composition), performance status tests, food log, urine color test, and other study assessments. These assessments will begin after cancer diagnosis but prior to intervention, and continue during treatment and at post-treatment visits.

DETAILED DESCRIPTION:
This is an observational, prospective device use study. 50 subjects will be enrolled in the study. The study will look at the changes in the participants body composition as they go through cancer treatment using the SOZO device. The SOZO device is intended to estimate the following body composition parameters: Fluid status (TBW, ECF, ICF), Total body composition (fat free mass, fat mass, % of weight), Metabolic report (active tissue mass, extracellular mass, basal metabolic rate), Skeletal muscle mass, Phase angle, Body mass index (BMI), Weight, and Hydration index (Hy-Dex) analysis. Participants will have 5 study visits during the course of their cancer treatment where SOZO measurements will be taken as well as other study measurements.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide consent
* Mentally and physically able to comply with protocol
* Age 18 and over
* Body Mass Index (BMI) ≤ 40 or body weight of <300 pounds
* Received first cancer diagnosis within 45 days of the Screening/Baseline study visit
* Diagnosis of cancer stage I-III
* Attempts to remove the cancer via chemotherapy, immunotherapy, radiation, etc. have not been initiated. Subjects will ideally enroll prior to any surgical cancer treatment, but enrollment post-surgery is allowable (capped at 15 subjects)
* Planned chemotherapy treatment not to exceed 6 months adjuvant treatment. Planned radiation and/or surgery, as well as planned maintenance therapy is allowable (i.e. continued treatment with endocrine therapy, monoclonal antibodies, or other longer-term treatments with minimal side effects) as determined by PI and approved by sponsor.

Exclusion Criteria:

* Active implanted medical device (cardiac pacemakers, defibrillators) or connected to electronic life support devices or patients with other metallic devices that would interfere with BIS measurements
* Amputees
* Any acute swelling condition diagnosed or actively being treated within 30 days of screening/baseline (including, but not limited to: acute heart failure, renal disease with dialysis, pulmonary edema, thrombophlebitis, deep vein thrombosis, pleural effusion, ascites, pregnancy)
* Patients with basal cell carcinoma or squamous cell skin cancer
* Currently suffering from uncontrolled intercurrent illness, including: ongoing/active infection, unstable angina pectoris, or cardiac arrhythmia
* Enrollment of female breast cancer patients not to exceed 60% of total projected enrollment. Once this threshold has been reached, these subjects will be excluded
* Planned orthopedic implant surgery
* Planned breast implant surgery
* Presence of or plan for breast expanders post-mastectomy
* Dependent upon transfusions
* Any history of organ transplant
* Presence of colostomy/ostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received their first diagnosis of any type of cancer stage I-III. Patients must have received this diagnosis within 45 days of the Screening/Baseline study visit. Patients will be ideally enrolled prior to surgical cancer treatment, but enrollment post-surgery is allowable.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
SOZO device can detect changes in body composition | Up to 6 months
  Assess change in body composition from baseline to final visit

SECONDARY OUTCOMES:
Correlate SOZO with 24-hour food recall. | Up to 6 months
  Assess correlation of SOZO measurements with 24-hour food recall.
Correlate SOZO with DEXA scan | Up to 6 months
  Assess correlation of SOZO measurements and DEXA scan (bone density with hip and spine measurements and whole body composition) results
Correlate SOZO with standard of care | Up to 6 months
  Assess correlation of SOZO measurements with standard of care measurements
Detect changes in physical performance | Up to 6 months
  Change from baseline in 6 minute walk test distance
Correlate SOZO with urine color test | Up to 6 months
  Assess correlation of SOZO measurements with urine color test.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Gluck, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health Cancer Institute Center for Integrative Oncology and Survivorship, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Churm D, Andrew IM, Holden K, Hildreth AJ, Hawkins C. A questionnaire study of the approach to the anorexia-cachexia syndrome in patients with cancer by staff in a district general hospital. Support Care Cancer. 2009 May;17(5):503-7. doi: 10.1007/s00520-008-0486-1. Epub 2008 Jul 29. PMID 18663481
- [Background] Spiro A, Baldwin C, Patterson A, Thomas J, Andreyev HJ. The views and practice of oncologists towards nutritional support in patients receiving chemotherapy. Br J Cancer. 2006 Aug 21;95(4):431-4. doi: 10.1038/sj.bjc.6603280. Epub 2006 Aug 1. PMID 16880793
- [Background] Pacelli F, Bossola M, Rosa F, Tortorelli AP, Papa V, Doglietto GB. Is malnutrition still a risk factor of postoperative complications in gastric cancer surgery? Clin Nutr. 2008 Jun;27(3):398-407. doi: 10.1016/j.clnu.2008.03.002. Epub 2008 Apr 23. PMID 18436350
- [Background] Bachmann J, Heiligensetzer M, Krakowski-Roosen H, Buchler MW, Friess H, Martignoni ME. Cachexia worsens prognosis in patients with resectable pancreatic cancer. J Gastrointest Surg. 2008 Jul;12(7):1193-201. doi: 10.1007/s11605-008-0505-z. Epub 2008 Mar 18. PMID 18347879
- [Background] Dewys WD, Begg C, Lavin PT, Band PR, Bennett JM, Bertino JR, Cohen MH, Douglass HO Jr, Engstrom PF, Ezdinli EZ, Horton J, Johnson GJ, Moertel CG, Oken MM, Perlia C, Rosenbaum C, Silverstein MN, Skeel RT, Sponzo RW, Tormey DC. Prognostic effect of weight loss prior to chemotherapy in cancer patients. Eastern Cooperative Oncology Group. Am J Med. 1980 Oct;69(4):491-7. doi: 10.1016/s0149-2918(05)80001-3. PMID 7424938
- [Background] Fearon KC, Voss AC, Hustead DS; Cancer Cachexia Study Group. Definition of cancer cachexia: effect of weight loss, reduced food intake, and systemic inflammation on functional status and prognosis. Am J Clin Nutr. 2006 Jun;83(6):1345-50. doi: 10.1093/ajcn/83.6.1345. PMID 16762946
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Tisdale MJ. Mechanisms of cancer cachexia. Physiol Rev. 2009 Apr;89(2):381-410. doi: 10.1152/physrev.00016.2008. PMID 19342610
- [Background] Strassmann G, Fong M, Kenney JS, Jacob CO. Evidence for the involvement of interleukin 6 in experimental cancer cachexia. J Clin Invest. 1992 May;89(5):1681-4. doi: 10.1172/JCI115767. PMID 1569207
- [Background] Falconer JS, Fearon KC, Ross JA, Elton R, Wigmore SJ, Garden OJ, Carter DC. Acute-phase protein response and survival duration of patients with pancreatic cancer. Cancer. 1995 Apr 15;75(8):2077-82. doi: 10.1002/1097-0142(19950415)75:83.0.co;2-9. PMID 7535184
- [Background] Terwee CB, Nieveen Van Dijkum EJ, Gouma DJ, Bakkevold KE, Klinkenbijl JH, Wade TP, van Wagensveld BA, Wong A, van der Meulen JH. Pooling of prognostic studies in cancer of the pancreatic head and periampullary region: the Triple-P study. Triple-P study group. Eur J Surg. 2000 Sep;166(9):706-12. doi: 10.1080/110241500750008466. PMID 11034467